CLINICAL TRIAL: NCT00558350
Title: Systemic, Intrapulmonary and Pleural Inflammatory Reaction in Patients Undergoing Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 68/07
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Lung Neoplasms
Keywords: lobectomy; inflammatory reaction; intrapulmonary; intrapleural
MeSH Terms: conditions — Lung Neoplasms; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: lobectomy / segmentectomy in patients with lung cancer

SUMMARY:
Inflammatory reaction in different compartments of the body may have a negative effect on outcome. This study assesses the inflammatory reaction systemically, intrapulmonary and intrapleural by measuring different cytokines. Patients with lung cancer undergoing lobectomy or segmentectomy are included in the study. Hypothesis: The inflammatory reaction in the pleural space is high compared to the systemic and intrapulmonary ones.

ELIGIBILITY:
Inclusion Criteria:

* elective lobectomy
* elective segmentectomy
* 20-90 years
* informed consent given

Exclusion Criteria:

* emergency operations
* pneumonectomy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients undergoing lobectomy or segmentectomy for lung cancer at a single institution
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2007-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Cytokine levels in blood, bronchial lavage fluid and pleural fluid | 2 years
Correlation between cytokine levels and pulmonary morbidity | 2 years

SECONDARY OUTCOMES:
Comparison of this collective with transthoracic esophagectomies and evaluation of the inflammatory reactions (esophageal collective registered:NCT00512265) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Urs Zingg, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland